CLINICAL TRIAL: NCT03902743
Title: Anticipatory Care Planning Intervention for Older Adults at Risk of Functional Decline: A Primary Care Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University, Belfast (Other)
Collaborators: Royal College of Surgeons, Ireland (Other); National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Kevin Brazil, Professor Kevin Brazil, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B18/46
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive an Anticipatory Care Plan
  Interventions: Other: Anticipatory Care Plan group
- Control group (No Intervention): Usual care

INTERVENTIONS:
Other: Anticipatory Care Plan group — The Anticipatory Care Plan will be delivered by a trained nurse. At the initial visit, the nurse will conduct a hollistic assessment using the EasyCare Assessment Tool. Following this visit, the nurse will draft a strucutred summary report of the home visit to include patient goals, preferences for care, identified problems and action list. The nurse will then consult with a pharmacist to identify any potential inappropriate prescribing. The nurse will then meet with the participants GP and review and provide feedback. The nurse will then re visit participants and discuss the report and agree a support plan and actions for follow up.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to explore the feasibility of delivering anticipatory care planning provided by nurses through a series of home visits. Many people with long-term health conditions can benefit from an anticipatory care plan as it helps them feel more in control of their life and allows them to manage changes in their health and well-being. The purpose of this study is to find out if effect of home visits by specially trained nurses for people aged 70 years and over who have been identified as being 'at risk' of developing frailty would be beneficial. Half of the patients in this study will receive home visits from trained nurses in addition to their usual care. Nurses will work with their GP, other healthcare providers and possibly family caregivers to plan and arrange any additional services that the participants require. The other half of patients in the study will receive usual care.

DETAILED DESCRIPTION:
Aim: to determine the feasibility of a cluster randomised trial to evaluate the implementation and outcomes of Anticipatory Care Planning (ACP) in primary care to assist older adults identified as at risk for functional decline by developing a personalised support plan.

Design and sample:

We will perform a feasibility cluster randomised controlled trial where 8 primary care practises will be randomly assigned (4 facilities per arm) to the intervention group versus usual care alone. Randomisation will be stratified according to location (Northern Ireland /Republic of Ireland - Louth, Monaghan). Primary care practices will be randomly allocated to the intervention or usual care arm before patient screening for risk of functional decline. A total of 64 patients (32 per study arm, 8 patients, randomly selected, per primary care practise) will be enrolled into the study. A sample of 32 patients per study arm is considered adequate to allow the size of any definitive trial to be determined more accurately and therefore minimise the number of patients required overall.

Setting:

Practices located in Northern Ireland will be recruited via the Northern Ireland Clinical Research Network (Primary Care). In the Republic of Ireland the HRB Primary Care Trials Network will recruit primary care practises located in the border counties of Louth and Monaghan. Practises will be drawn from both urban and rural settings that serve a socioeconomically deprived population.

Patient enrolment:

Individuals who screen as at risk of functional decline will be sent a letter from their GP inviting them to participate in the study. A project research assistant will recruit consenting patients by telephone. Allocation to the intervention vs. usual care will be communicated to the study participant by a member of the research team after the research assistant has obtained consent and conducted the baseline-standardised interview. In the case of two or more eligible participants in any one household, all will be eligible for enrolment into the study. In the intervention arm the study nurse employed by the project will then commence arrangements to visit the appropriate patients.

Intervention:

The nurse led ACP intervention will be integrated into regular care where the study nurse will involve the patients' GP in care planning and is informed about patients' goals and plans. As a first step in the intervention, the study nurse will contact the patient by telephone to schedule an initial home visit. This will typically be conducted within 4 weeks of the return of the participant's PRISMA 7 postal questionnaire. At the initial home visit the study nurse will, with the aid of a medical summary including current repeat prescription provided by the GP practise, will employ a structured protocol conduct a brief Comprehensive Geriatric Assessment (CGA) that will also encourage discussion about present and future care and patient goals.

Following the initial home visit the study nurse will draft a structured summary report of the home visit that will include patient goals, preferences for care, identified problems and action list. The study nurse will forward to a pharmacist, who will be an adjunct to the study, the summary report generated from the brief CGA highlighting the patient medication list and the identification of potentially inappropriate prescribing (PIP). The pharmacist will cross check and verify the presence of PIPs. A record will be maintained by the pharmacist on the accuracy of the study nurse identifying PIPs during the trial. The results of this audit will contribute to the finalisation of the intervention. Subsequent to PIP feedback from the pharmacist the study nurse will finalize the summary report and will meet with the GP who will be informed through a structured format patients goals and wishes, results of the patient assessment, problem list and recommended actions. The GP with appropriate participation of other members of the health care team, will review, provide feedback and confirm agreement with the plan of care.

In the second home visit the study nurse will meet with the patient and family carer to discuss identified problems, review proposed options for support, document the agreed support plan and consider options for follow up and set a date for review. The study nurse may conduct, depending on clinical need, the second visit in the patients' home or the GP practise so the GP can be present. The finalised care plan will be left with the patient and a copy will be placed in the patient's chart in the GP practise.

All outcome measures will be assessed at baseline, six weeks and six months.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥70 years
* In receipt of a valid general medical services (GMS) card in the Republic of Ireland, or for Northern Ireland registered for NHS primary care services
* ability to complete a postal questionnaire

Exclusion Criteria:

* receiving specialist palliative care
* record of assessed cognitive impairment at the level that would impact their ability to complete screening postal questionnaire, outcome measures and participate in a patient care conference(s) (defined as Mini Mental State Examination (MMSE) ≤20)
* experiencing a psychotic episode at the time of recruitment
* hospitalised long-term, in a nursing home, homeless or in sheltered accommodation

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
EQ-5D-5L | 10 minutes
  Is a widely used self-reported generic measure of health reported quality of life that has been validated in different patient populations. The five-level version contains the same dimensions as the earlier three-level version but has been designed to provide greater reliability and sensitivity.
Center for Epidemiological Studies Depression Scale (CES-D) | 10 minutes
  This 20- item scale has been used extensively with older adults. Respondents use a four choice scale to rate how they have felt in the past week expressing depressed mood.

SECONDARY OUTCOMES:
Patient Assessment of Chronic Illness Care (PACIC) Scale | 15 minutes
  This 20 item scale was designed to assess from the patient perspective the receipt of patient-centered care and self-management behaviors.
Health Economic Evaluation | 15 minutes
  The health economic analysis will consist of trial-based economic evaluation and will incorporate both cost effectiveness analysis and cost utility analysis to compare the alternative treatment strategies: (1) the Anticipatory Care Planning (ACP) Intervention; and (2) usual care in general practice.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Brazil, PhD, Principal Investigator — Queens University Belfast
Locations (1):
- Queens University Belfast, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Plan in preparation
Supporting Information: Study Protocol
Time Frame: August 2021
Access Criteria: Those requesting access will be required to submit a letter of intent to the study PI after which the research team will review their request

REFERENCES:
- [Derived] Brazil K, Cardwell C, Carter G, Clarke M, Corry DAS, Fahey T, Gillespie P, Hobbins A, McGlade K, O'Halloran P, O'Neill N, Wallace E, Doyle F. Anticipatory care planning for community-dwelling older adults at risk of functional decline: a feasibility cluster randomized controlled trial. BMC Geriatr. 2022 May 25;22(1):452. doi: 10.1186/s12877-022-03128-x. PMID 35610581
- [Derived] Corry DAS, Carter G, Doyle F, Fahey T, Gillespie P, McGlade K, O'Halloran P, O'Neill N, Wallace E, Brazil K. Successful implementation of a trans-jurisdictional, primary care, anticipatory care planning intervention for older adults at risk of functional decline: interviews with key health professionals. BMC Health Serv Res. 2021 Aug 25;21(1):871. doi: 10.1186/s12913-021-06896-1. PMID 34433441
- [Derived] Brazil K, Scott D, Wallace E, Clarke M, Fahey T, Gillespie P, O'Halloran P, Cardwell C, Carter G, McGlade K, Doyle F. Anticipatory care planning intervention for older adults at risk of functional decline: study protocol for a primary care cluster feasibility randomised trial. Trials. 2020 Feb 11;21(1):168. doi: 10.1186/s13063-020-4100-2. PMID 32046767

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT03902743/Prot_SAP_000.pdf